CLINICAL TRIAL: NCT07283510
Title: Exploring the Effects of a Community-based Functional Fitness Program on Physical Function Among Adults Aging With Mobility Disability: A Pilot Study
Brief Title: Community-based Functional Fitness for Adults Aging With Mobility Disability
Acronym: AAIMLCOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Lyndsie Koon, Assistant Research Professor, University of Kansas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GR17636
Record Dates: First submitted 2025-04-15; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Mobility Disability; Older Adults
Keywords: Functional Fitness; Mobility Disability; Aging with Disability; Older Adults; Community-based Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-person Functional Fitness Arm (Experimental): In-person, thrice weekly, 16-week functional fitness arm took place at community-based functional fitness affiliate locations
  Interventions: Behavioral: Functional Fitness

INTERVENTIONS:
Behavioral: Functional Fitness — Location/availability: To increase access, FF sessions will be available at 3 facilities located in the greater Kansas City area. Each facility has accessible space, equipment, and certified Adaptive and Inclusive FF trainers to deliver the intervention. Sessions will be capped at 10 participants and led by a minimum of two certified trainers. Acclimation: Prior to initiating the intervention, participants will complete two acclimation sessions to learn the basic FF movements adapted to their abilities and required safety protocols. FF session frequency: Participants will be asked to attend 3 - 60 min. group sessions/wk. over 16 wks. (48 total sessions). FF session content: Each session will include a warm-up (~15 min.) FF (~30 min) and a cool down (~15 min). Sessions will be standardized; however, all aspects of the session (movements, load) will be adapted to individual capabilities. FF prescriptions for each session and participant adaptations will be documented

SUMMARY:
Evaluate the feasibility and potential effectiveness of a 12-week, high-intensity functional training (HIFT) intervention on frailty in older adults (60+) with mobility disabilities (MD) who are ambulatory

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine the feasibility and effectiveness of an adaptive and inclusive community-based exercise intervention targeting parameters associated with the development of frailty in older adults with a mobility disability (MD). Adults aging with MD differ from those aging into MD, as this population is managing an original disability acquired earlier in life with secondary conditions, in addition to age-related changes. The interactive effects of aging and disability may result in greater susceptibility to frailty, defined as a state of vulnerability that increases risk for adverse health outcomes. Exercise is a potentially viable option for supporting functional health factors that contribute to frailty, as exercise participation has been associated with improvements in multiple functional outcomes (e.g., balance, strength) among people with MD, to a greater extent than other health outcomes (e.g., mental, metabolic health). Many exercise trials demonstrating promising results are conducted in laboratory or clinical settings, where long-term participation is often unsustainable and transferability to community settings is limited. Therefore, the investigators propose to evaluate the feasibility and effects of a community-based, adaptable, and inclusive exercise program known as Functional Fitness (FF) for adults aging with MD. FF is one of the fastest-growing fitness trends and incorporates movement patterns that simulate everyday activities important for individuals with MD, including transferring, picking up an object from a seated position, and ambulating without supports.

The investigators will conduct a single-arm pilot trial of a 16-week community-based Functional Fitness (FF) intervention (three 60-minute sessions per week) in 12 older adults (aged 60 years and older) with a permanent mobility disability. The study will address the following aims:

Aim 1. Feasibility of the FF intervention will be assessed based on participant recruitment, session attendance, retention, and completion of all outcome assessments. Semi-structured exit interviews will be conducted with all participants to elicit feedback on suggested intervention improvements, perceptions of intervention length and frequency, satisfaction with instructors, exercise facilities, and session content, as well as challenges related to intervention compliance.

Aim 2. Effectiveness of the 16-week intervention will be evaluated based on changes in functional outcomes independently associated with frailty, including mobility, balance, strength, and psychosocial outcomes. FF will be implemented through an existing community program (Adaptive Athletes in Motion) that has served the disability community for more than five years by providing scholarship-based Functional Fitness programming to individuals with a range of disability types, primarily mobility-related disabilities. Given its prevalence and inclusive design, FF provides a framework for widespread adoption, implementation, and maintenance of exercise programming for older adults with MD. Results from the proposed trial will generate preliminary evidence regarding the feasibility of FF for adults aging with MD and provide novel empirical data on the program's potential effects on frailty-related outcomes in an understudied population at increased risk for loss of functional independence due to the intersection of aging and disability.

ELIGIBILITY:
Inclusion Criteria:

Aged 60 years or older

Presence of a permanent mobility disability (duration of at least 1 year)

Ambulatory (does not use a manual or power wheelchair for mobility)

Not currently participating in a structured exercise program

No significant health impairment that would contraindicate participation in Functional Fitness, as confirmed by a primary care provider

Ability to serve as one's own guardian and provide informed consent

Exclusion Criteria:

Inability to utilize reliable transportation to travel to and from the fitness facility three times per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Walking Speed as Assessed by the 10-Meter Walk Test (m/s) | From enrollment to the end of the intervention at 16-weeks
  Walking speed will be assessed using the 10-meter walk test. Participants will be instructed to walk a marked 10-meter distance at a comfortable pace. Walking speed will be calculated in meters per second, with higher values indicating faster walking speed and better mobility.
Change in Aerobic Endurance as Assessed by the 2-Minute Step Test (steps) | From enrollment to the end of treatment at 16-weeks
  Aerobic endurance will be assessed using the 2-minute step test. The total number of steps completed within two minutes will be recorded, with higher step counts indicating greater aerobic endurance.
Change in Functional Mobility as Assessed by the Timed Up and Go Test (seconds) | From enrollment to the end of treatment at 16-weeks
  Functional mobility will be assessed using the Timed Up and Go test. Time (in seconds) required to stand from a seated position, walk a standardized distance, turn, return, and sit will be recorded. Shorter completion times indicate better functional mobility.
Change in Lower Extremity Functional Strength as Assessed by the Five Times Sit-to-Stand Test (seconds) | From enrollment to the end of treatment at 16-weeks
  Lower extremity functional strength will be assessed using the Five Times Sit-to-Stand test. Time (in seconds) required to complete five repeated sit-to-stand transitions will be recorded, with shorter times indicating greater functional strength.

SECONDARY OUTCOMES:
Change in Balance as Assessed by the Berg Balance Scale (score) | From enrollment to the end of treatment at 16-weeks
  Balance will be assessed using the Berg Balance Scale, a 14-item performance-based measure of static and dynamic balance. Total scores range from 0 to 56, with higher scores indicating better balance performance.
Change in Postural Stability as Assessed by Postural Sway Measures (center of pressure displacement) | From enrollment to the end of treatment at 16-weeks
  Postural stability will be assessed by quantifying postural sway during quiet standing. Measures will include displacement of the center of pressure over a fixed period, with greater sway (in degrees) indicating poorer postural stability.
Change in Handgrip Strength as Assessed by Jamar Smart Digital Hand Dynamometry (kg) | From enrollment to the end of treatment at 16-weeks
  Grip strength of both the dominant and non-dominant hands will be assessed using a Jamar Smart Digital hand dynamometer. Peak grip force will be recorded in kilograms, with higher values indicating greater upper extremity strength.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are still evaluating the feasibility of sharing individual participant data (IPD) based on privacy considerations, data use agreements, and input from our institutional review board. We recognize the value of data sharing for advancing research and plan to assess appropriate mechanisms to ensure responsible access to de-identified IPD, if permitted.